CLINICAL TRIAL: NCT05435300
Title: Does tDCS Change Synaptic Density in the Brains of Patients With Schizophrenia
Status: Recruiting | Type: Observational
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Sponsor
Other Study IDs: 118/2020
Record Dates: First submitted 2022-06-23; First posted 2022-06-28 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-03

CONDITIONS: Schizophrenia; Schizoaffective
Keywords: Positron emission tomography
MeSH Terms: conditions — Schizophrenia | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Schizophrenia/Schizoaffective Disorder: Participants with Schizophrenia/Schizoaffective Disorder and currently enrolled in the tDCS-adherence parent study (REB# 103-2018).
  Interventions: Other: PET Scan

INTERVENTIONS:
Other: PET Scan — Participants will undergo two PET scans throughout the study.

SUMMARY:
This study will examine changes in synaptic density with transcranial direct current stimulation (tDCS) in the brains of patients with schizophrenia. Synaptic density levels will be measured using a novel positron emission tomography (PET) radiotracer [18F]SDM-8, which is currently the best-in-class method to quantify synaptic density in humans. This will be a companion study to a parent study by our group examining the effects of tDCS on treatment adherence in schizophrenia (REB #103-2018).

DETAILED DESCRIPTION:
The aim of our study is to examine if tDCS induces synaptic density changes in patients with schizophrenia using [18F]SDM-8. Our study will help elucidate the mechanism through which tDCS affects the brain.

PET scans will be offered to participants that meet the inclusion and exclusion criteria at the initial screening visit. Participants will be scanned with the novel PET tracer [18F]SDM-8 to quantify synaptic density levels. PET scans will be timed to coincide to the two time-points, before and after 2-weeks of tDCS treatment that is completed under the parent study protocol (REB #103-2018). Clinical assessments will be done at the same time.

ELIGIBILITY:
Inclusion Criteria:

Enrolment in the tDCS-adherence parent study (REB# 103-2018). The parent study inclusion criteria are:

1. Male or female participants of any race or ethnicity
2. Inpatients or outpatients ≥18 years of age
3. DSM-V diagnosis of schizophrenia or schizoaffective disorder
4. Capable of consenting to participate in the research study
5. On a stable dose of oral antipsychotic drug and other concomitant medications for at least 2 months, and unlikely to undergo changes in dose during the study.

Exclusion Criteria:

The exclusion criteria for this study will be the same as the parent study (REB 103-2018). The parent study exclusion criteria are:

1. Unwilling or incapable to consent to the study based on the MacArthur Test of Competence
2. Unstable medical or any concomitant major medical or neurological illness, including a history of seizures
3. Acute suicidal or homicidal ideation
4. Formal thought disorder rating ≥3 on the Positive and Negative Syndrome Scale (PANSS) P2 conceptual disorganization item
5. DSM-V substance dependence (except caffeine, nicotine, and cannabis/marijuana) within 1 month of entering the study
6. Positive urine drug screen except for cannabis/marijuana at the screening visit
7. Metal implants or pacemaker precluding an MRI scan or other contraindications to MRI (e.g., claustrophobia)
8. Pregnancy
9. Score <32 on the Wide Range Achievement Test-III

Additional exclusion criteria for this companion study are:

1. Unwilling or incapable to consent to the study based on the MacArthur Test of Competence
2. Exposure to long-acting injectable antipsychotics in the last 6 months
3. Exceeding allowed annual radiation exposure levels (20 mSv), as outlined by our PET Centre guidelines
4. Receiving treatment with medications such as levetiracetam that blocks SV2a binding
5. Disorders of coagulation or taking anticoagulant medication
6. Having completed multiple PET scans in the past, such that participation in this study would cause participant to exceed lifetime limit (8 PET scans)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will have Schizophrenia/Schizoaffective Disorder and currently enrolled in the tDCS-adherence parent study (REB# 103-2018).
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-09-17 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Synaptic density changes | PET scans will be timed to coincide to the two time-points, before and after 2-weeks of tDCS treatment that is completed under the parent study protocol (REB #103-2018)
  The primary outcome measure is the [18F]SDM-8 standard uptake value (SUV) and distribution volume ratio (DVR) in cortical and subcortical gray matter regions, measured by PET Scans

CONTACTS AND LOCATIONS:
Overall Officials: Philip Gerretsen, MD, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Centre for Addiction and Mental Health (CAMH) is the leading mental health and addictions research facility in Canada, and one of the largest in the world. — https://www.camh.ca/en/science-and-research